CLINICAL TRIAL: NCT01326507
Title: Performances de l'h-FABP Pour Identifier dès Les Urgences Les Embolies Pulmonaires d'évolution défavorable
Brief Title: Prognostic Value of Heart-type Fatty Acid-Binding Protein (h-FABP) in Acute Pulmonary Embolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0900303; 2009-A00441-56 (Other: Afssaps)
Record Dates: First submitted 2009-11-06; First posted 2011-03-31 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Pulmonary Embolism
Keywords: pulmonary embolism; Heart-type fatty acid-binding protein; cardiac biomarkers; risk stratification
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Dosage de l'h-FABP — Dosage de l'h-FABP

SUMMARY:
The patients presenting with acute pulmonary embolism and right ventricular dysfunction are at high risk for life-threatening events and must be identified in the emergency department for adequate care and hospital admission. Echocardiography can identify right ventricular dysfunction, but this test is not always available, and echocardiographic criteria of right ventricular dysfunction vary among published studies. The primary purpose of this protocol is to study the prognostic value of a cardiac biomarker, h-FABP (heart-type Fatty Acid-Binding Protein) , to identify in the emergency department the patients presenting with high risk pulmonary embolism. As secondary outcomes, H-FABP results will be compared to other cardiac biomarkers (BNP, troponin) and clinical score performances that have been previously studied to stratify the prognosis of patients with pulmonary embolism in the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* patients with acute pulmonary embolism diagnosed in the emergency departement

Exclusion Criteria:

* patient under guardianship
* patient without social insurance
* pregnant women
* refusal to sign the consent
* myocardial infarction in the 10 days before pulmonary embolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2009-09; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
number of death by pulmonary embolism | 1 month
life-threatening pulmonary embolism (cardiopulmonary arrest, shock, mechanical ventilation) | 1 month
recurrent episode of pulmonary embolism | 1 month

SECONDARY OUTCOMES:
prognostic value of a clinical score (PESI), BNP and troponin in acute pulmonary embolism | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Dominique LAUQUE, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Hôpital Rangueil Service des urgences, Toulouse, France

REFERENCES:
- [Result] Lauque D, Maupas-Schwalm F, Bounes V, Juchet H, Bongard V, Roshdy A, Botella JM, Charpentier S. Predictive value of the heart-type fatty acid-binding protein and the Pulmonary Embolism Severity Index in patients with acute pulmonary embolism in the emergency department. Acad Emerg Med. 2014 Oct;21(10):1143-50. doi: 10.1111/acem.12484. PMID 25308138